CLINICAL TRIAL: NCT00003056
Title: Peripheral Blood Stem Cell Transplantation in Patients With Advanced Malignancies Eligible for Allogeneic Transplantation From Matched Related Donors: A Randomized Study of Cyclosporine/Methotrexate or Cyclosporine/T-Cell Depletion (CD34 Cell Selection) for GVHD Prophylaxis
Brief Title: Prevention of Graft-Versus-Host Disease in Patients With Advanced Leukemia or Lymphoma Who Are Eligible for Peripheral Stem Cell Transplantation
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Interim analysis indicated study should be terminated
Sponsor: Baxalta now part of Shire (Industry)
Responsible Party: Sponsor
Organization: Takeda (Industry)
Allocation: Randomized | Model: Parallel | Purpose: Supportive Care
Other Study IDs: BAXTER-302302; MCV-CCHR-9703-2A; CDR0000065709 (Registry Identifier: PDQ (Physician Data Query)); NCI-G97-1311
Record Dates: First submitted 1999-11-01; First posted 2004-05-24 (Estimated); Last update posted 2021-05-06 (Actual); Status verified 2021-05

CONDITIONS: Leukemia; Lymphoma; Graft Versus Host Disease
Keywords: recurrent adult diffuse small cleaved cell lymphoma; adult acute myeloid leukemia in remission; recurrent grade 2 follicular lymphoma; accelerated phase chronic myelogenous leukemia; adult acute lymphoblastic leukemia in remission; recurrent grade 1 follicular lymphoma; recurrent adult lymphoblastic lymphoma; recurrent marginal zone lymphoma; chronic phase chronic myelogenous leukemia; recurrent small lymphocytic lymphoma; recurrent grade 3 follicular lymphoma; recurrent adult Hodgkin lymphoma; recurrent adult acute lymphoblastic leukemia; recurrent adult immunoblastic large cell lymphoma; graft versus host disease; recurrent adult diffuse mixed cell lymphoma; recurrent mantle cell lymphoma; splenic marginal zone lymphoma; recurrent adult acute myeloid leukemia; extranodal marginal zone B-cell lymphoma of mucosa-associated lymphoid tissue; recurrent adult diffuse large cell lymphoma; nodal marginal zone B-cell lymphoma; recurrent adult Burkitt lymphoma
MeSH Terms: conditions — Leukemia; Lymphoma; Graft vs Host Disease; Lymphoma, Non-Hodgkin; Lymphoma, Follicular; Leukemia, Myeloid, Accelerated Phase; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Lymphoma, B-Cell, Marginal Zone; Leukemia, Myeloid, Chronic-Phase; Leukemia, Lymphocytic, Chronic, B-Cell; Hodgkin Disease; Lymphoma, Large-Cell, Immunoblastic; Lymphoma, Mantle-Cell; Leukemia, Myeloid, Acute; Lymphoma, Large B-Cell, Diffuse; Burkitt Lymphoma | interventions — Cyclosporine; Methotrexate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Unselected peripheral blood haemopoietic stem cells (PBSC) (Active Comparator): Unselected PBSC together with control graft versus host disease (GVHD) prophylaxis - Control
  Interventions: Drug: cyclosporine and methotrexate
- CD34+ cells isolated from PBSC (Experimental): CD34+ cells isolated from PBSC using the Isolex 300i system together with cyclosporine
  Interventions: Drug: cyclosporine

INTERVENTIONS:
Drug: cyclosporine
  Arms: CD34+ cells isolated from PBSC
Drug: cyclosporine and methotrexate
  Arms: Unselected peripheral blood haemopoietic stem cells (PBSC)

SUMMARY:
RATIONALE: Peripheral stem cell transplantation may be able to replace immune cells that were destroyed by chemotherapy or radiation therapy used to kill tumor cells. Sometimes the transplanted cells can make an immune response against the body's normal tissues.

PURPOSE: Randomized phase III trial to compare the effectiveness of cyclosporine plus methotrexate with cyclosporine plus T cell depletion for prevention of graft-versus-host disease during peripheral stem cell transplantation in patients who have advanced leukemia or lymphoma who are eligible for transplanted peripheral stem cells from a donor.

DETAILED DESCRIPTION:
OBJECTIVES: I. Demonstrate that the graft versus host disease (GVHD) prophylactic regimen consisting of T-cell depletion and cyclosporine results in less toxicity than the control regimen of methotrexate and cyclosporine in recipients of peripheral blood stem cell transplants. II. Monitor safety of the two regimens in order to assure that the treatment regimen dose not result in any increase in serious or unexpected toxicities, does not compromise the efficacy of GVHD prophylaxis, and does not compromise the efficacy of the disease therapy.

OUTLINE: This is a multicenter, controlled, randomized trial. Patients are assigned to high or low risk groups and randomized to the control or treatment arms. Patients are stratified by risk group and by site. Mobilization, apheresis, and successful cryopreservation of the minimum number of CD34 cells for transplant has to be achieved prior to initiating cytoreductive therapy. Following intensive cytoreductive therapy, patients receive either unselected peripheral blood stem cells (PBSC) together with the control graft versus host disease (GVHD) prophylaxis regimen or CD34+ cells isolated from PBSC with cyclosporine. In the control group, GVHD prophylaxis consists of two drug therapies, cyclosporine and methotrexate. The cyclosporine is administered first by IV continuous infusion and then later orally, twice a day, in decreasing increments for 180 days. Methotrexate is administered by IV on days 1, 3, 6, and 11. Cyclosporine is discontinued after day +180 if there is no evidence of GVHD. In the treatment group, GVHD prophylaxis consists of T cell depletion of the transplant product using the Isolex positive selection procedure (Isolex selected CD34+ cells) and cyclosporine. The cyclosporine is administered at the same doses and increments as in the control group. In cases where there still is acute or chronic GVHD, the patient is given the appropriate salvage regimens. Patients are followed monthly for 6 months after transplant, and then for 2 years to monitor relapses.

PROJECTED ACCRUAL: There will be 200 patients accrued (100 in each arm) in this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS: - Acute lymphocytic leukemia (ALL) with documented chemosensitivity (complete response [CR], partial response [PR], or minor response [MR]) in first or second remission, first or second relapse, or high risk ALL with Ph positive 9/22 translocation; OR - Acute myelogenous leukemia (AML) with documented chemosensitivity (CR, PR, or MR) in first or second remission, or first or second relapse; OR - Chronic myelogenous leukemia (CML), chronic or accelerated, that is not in blast crisis; OR - Hodgkin's disease or non-Hodgkin's lymphoma with documented chemosensitivity in first or second relapse Consenting human lymphocyte antigen (HLA)-identical related donor required No active central nervous system (CNS) or skin leukemia involvement No disease that requires additional mediastinal radiation

PATIENT CHARACTERISTICS: Age: 18-55 Performance status: Karnofsky 70-100% Life expectancy: Greater than 8 weeks Hematopoietic: Not specified Hepatic: Bilirubin less than 1.5 times normal serum glutamate oxalo-acetate transaminase (SGOT) less than 2 times normal Renal: Creatinine less than 1.5 times normal Cardiovascular: Left ventricular ejection fraction at rest at least 40% or within normal range Pulmonary: diffusing capacity of the lung for carbon monoxide (DLCO) greater than 45% of predicted or within normal range Other: HIV negative At least 2 weeks since any active infection requiring intravenous treatment with antifungal, antibacterial or antiviral agents with the exception of coagulase negative staphylococcal line infection No coexisting medical problems that would significantly increase the risk of the transplant procedure Not pregnant or nursing

PRIOR CONCURRENT THERAPY: No more that 2 prior therapy regimens Biologic therapy: No prior autologous or allogeneic bone marrow or peripheral blood stem cell transplant Chemotherapy: Not specified Endocrine therapy: Not specified Radiotherapy: Prior radiation therapy subject to dose requirements Surgery: Not specified Other: At least 2 weeks since intravenous treatment with antifungal, antibacterial or antiviral agents, except for treatment of coagulase negative staphylococcal infection of an IV or central line

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 105 (Actual)
Dates: Start 1997-04-01 (Actual); Primary Completion 2003-06-01 (Actual); Study Completion 2003-06-01 (Actual)

PRIMARY OUTCOMES:
Time to neutrophil engraftment | Month 1, post-transplant
Time to neutrophil engraftment | Month 2, post-transplant
Time to neutrophil engraftment | Month 3, post-transplant
Time to neutrophil engraftment | Month 4, post-transplant
Time to neutrophil engraftment | Month 5, post-transplant
Time to neutrophil engraftment | Month 6, post-transplant

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda
Locations (13):
- United States (12):
  - Los Angeles, California
  - Jacksonville, Florida
  - Atlanta, Georgia
  - Indianapolis, Indiana
  - Lawrence, Kansas
  - Saint Paul, Minnesota
  - Kansas City, Missouri
  - St Louis, Missouri
  - Hackensack, New Jersey
  - Pittsburgh, Pennsylvania
  - San Antonio, Texas
  - Richmond, Virginia
- Adelaide, South Australia, Australia